CLINICAL TRIAL: NCT01949935
Title: MIR-CABG: A Randomized, Double-blind, Placebo-controlled, Single-Center Study to Evaluate the Impact of Mupirocin on Infection Rate Post Coronary Artery Bypass Grafting
Brief Title: Efficacy Study of Mupirocin on Infection After Coronary Artery Bypass Grafting
Acronym: MIR-CABG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Horizon Health Network (Other)
Responsible Party: Principal Investigator, Dr Craig Brown, Director of Clinical Trials, New Brunswick Heart Centre, Horizon Health Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NBHC-MIR004
Record Dates: First submitted 2012-12-05; First posted 2013-09-25 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Surgical Site Infections
Keywords: Mupirocin; Surgical Site Infections; Coronary Artery Bypass Grafting
MeSH Terms: conditions — Surgical Wound Infection | interventions — Mupirocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Placebo made from Glaxal base Applied once 1 day preoperatively and bid for 3 days postoperatively.
  Interventions: Drug: Mupirocin
- Mupirocin (Experimental): Mupirocin ointment applied to nares once 1 day preoperatively and bid for 3 days postoperatively.
  Interventions: Drug: Mupirocin

INTERVENTIONS:
Drug: Mupirocin
  Other Names: Bactroban

SUMMARY:
The hypothesis is that application of Mupirocin to the nose before and after coronary artery bypass grafting surgery will reduce the incidence of surgical site infections.

DETAILED DESCRIPTION:
Mupirocin applied to the nares is effective in eradicating nasal carriage of Staphylococcus species. Abundant evidence has documented that a majority of gram positive surgical site infections share bacterial phenotypes identical with nasal phage types. Conflicting literature exists regarding the efficacy of mupirocin in reducing the incidence of surgical site infections. A randomized prospective double-blind placebo-controlled trial is needed to help settle this question in the setting of coronary artery bypass grafting surgery where surgical site infections carry significant morbidity, cost, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years old undergoing Coronary Artery Bypass Grafting Surgery (CABG) with or without concomitant cardiac valve surgery or other cardiac surgery,
* Median sternotomy wound
* Capable of informed consent

Exclusion Criteria:

* Allergy to mupirocin or components
* Pregnant or lactating females
* Emergency surgery
* Pre-existing ongoing infection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 974 (Actual)
Dates: Start 2009-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection | <30 days post operation
  Surgical site infections (SSI) are classified as superficial, deep, or organ surgical site infections based on CDC definition.

SECONDARY OUTCOMES:
Mortality | < or = 30 days post operation
Serious adverse durg effects | < or = 30 day post operation
  Rashes, rhinorrhea, pruritis, bleeding from nares
S. aureus carrier status | < or = 30 day post operation
  Nasal carriage of Staphylococcus aureus assess pre-intervention and post-intervention.

OTHER OUTCOMES:
Incidence of subtypes of surgical site infections. | < or = 30 days post operation.
  Subtypes include deep sternal wound, mediastinitis, leg saphenous vein harvest site infections.
Incidence of pneumonia | < or = 30 days post operation.
  As diagnosed by sputum, radiographic, and clinical means.

CONTACTS AND LOCATIONS:
Overall Officials: Craig D Brown, BSc (Med), MD, FRCSC, FACS, Principal Investigator — New Brunswick Heart Centre
Locations (1):
- New Brunswick Heart Centre, Saint John Regional Hospital, Saint John, New Brunswick, Canada